CLINICAL TRIAL: NCT04736264
Title: Malay Glaucoma Eye Study II: Elucidating Navigation, Mobility and Reading Ability to Improve Quality of Life and Progression of Primary Glaucoma
Brief Title: Malay Glaucoma Eye Study II Navigation, Mobility and Reading Ability in Primary Glaucoma
Acronym: MaGESII
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universiti Sains Malaysia (Other)
Collaborators: Ministry of Health, Malaysia (Other Government); Universiti Teknologi Mara (Other)
Responsible Party: Principal Investigator, Liza Sharmini Ahmad Tajudin, Professor, Head of Glaucoma Research, Principal Investigator, Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Universiti Sains Malaysia; RUI 1001/PPSP/8012350 (Other Grant/Funding Number: Universiti Sains Malaysia)
Record Dates: First submitted 2020-11-28; First posted 2021-02-03 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Primary Open Angle Glaucoma; Primary Angle Closure Glaucoma
Keywords: Rehabilitation; Navigation; Mobility; Physical activity; Reading; Quality of life; Oxidative Stress; Exercise
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma, Angle-Closure; Motor Activity | interventions — Range of Motion, Articular

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rehabilitation group (Active Comparator): This is the phase 3 of the entire research protocol. Phase 3 will be initiated once the phase 2 (development of rehabilitation module) is completed. A user friendly and inexpensive device and program with minimal usage of low vision aid will be designed and piloted. There are 3 different rehabilitation modules.
  A total of 300 primary glaucoma patients will be recruited and randomized using SNOSE: 150 intervention group and 150 non-intervention group. The intervention group will comprised of 150 primary glaucoma patients who will be assigned to different rehabilitation program:
  1. navigation and mobility (50 patients)
  2. physical activities including special exercise (50 patients)
  3. reading (50 patients) There will be no patient who will be involved in more than one rehabilitation program at anytime.
  Interventions: Other: Visual rehabilitation module: navigation and mobility; Other: Visual rehabilitation module: exercise; Other: Visual rehabilitation module: reading
- Non-rehabilititation group (No Intervention): Group of primary glaucoma patients who are not taught and practiced the new rehabilitation module for navigation, physical activity (exercise) and reading. They will be asked to continue their regular activities and provided with the similar reading material (book) to read daily.

INTERVENTIONS:
Other: Visual rehabilitation module: navigation and mobility — The visual rehabilitation regime consist of education and activity include dressing, feeding, personal hygiene and grooming activities, functional mobility, room orientation and memory, reading, eye hand coordination and also optokinetic training programme. A diary will be given to assess their compliance. Reassessment based on the number of fall, stumble etc when they go through a maze (developed in Phase 1)will be done every 2weeks for 8 weeks (4 times), every 4 weeks for next 8 weeks (2 times) and the final assessment 8 weeks later. A total study intervention will be 24 weeks
  Arms: Rehabilitation group
Other: Visual rehabilitation module: exercise — An instruction course will be conducted and a CD (with step by step exercise demonstration) will be given to the patients in group A. They will be asked to come for another session in 2 weeks. Then they will be asked to conduct the exercise for at least three times a week for 24 weeks. Exercise diary and accelerometer will also be given to patients of both groups. They will be seen in the clinic every 8 weeks.
  Arms: Rehabilitation group
Other: Visual rehabilitation module: reading — Patient in intervention group will be asked to complete a reading task (reading the given book) a day, number of pages completed in an hour per day and time taken to complete a page in given book. They are asked to complete the books within 24 weeks with follow up every 8 weeks.
  Arms: Rehabilitation group

SUMMARY:
With the improvement of health system, the life span of Asians has increased tremendously especially in Malaysia. As an early preparation to be an 'aging country' in 2023, Malaysia needs to prepare infrastructure and policy to improve quality of life (QoL) in older adults. Glaucoma is an aging related chronic disease that cause progressive optic neuropathy and visual field defect1. The main aim of glaucoma treatment is to slow down disease progression and preserve patient's QoL2. Modification of intraocular (IOP) is believed to be the mainstay of treatment but may not prevent progression of the disease. Modification of lifestyle has been found to change the prognosis of many chronic diseases such as diabetes mellitus. However, there is minimal evidence on the effect of lifestyle modification on glaucoma. Although constricted visual field almost asymptomatic especially in primary open angle glaucoma but many domestic injuries such as fall has been reported. Glaucoma patients reported greatest restriction with mobility especially driving compared to the other domains3,4. Reduction of walking and moderate-to-vigorous physical activity was also found in those with bilateral visual field loss5. Progressive constriction of visual field has been found to increase dependency, reduce mobility, pleasure of reading and QoL of glaucoma patients6. This will lead to psychological and emotional disturbance, in certain cases even resulted in depression. On the other hand, being physically active is found to have some protective effect against development and severity of glaucoma8,9. Thus, identifying problems related to physical activities in constricted visual field is important for improvement of rehabilitation and exercise regime for glaucoma patients. An exercise regime must be effective without causing major changes to IOP, safe in patients with constricted visual field and sensitive to social culture of Malaysians. Addressing these issues will lessen dependency and promotes healthy living among older adults. Improvement in navigation perhaps may increase the physical activities in glaucoma. Reading is another important pleasure in life. Visual field defect in glaucoma patients has been reported to associate with slower reading speed, saccade rate and visual span10,11. Identification of factors associated with difficulty in reading among glaucoma patients and development of rehabilitation regime in reading may improve the happiness index in literate patients. Nevertheless, there is no specific rehabilitation program to improve reading abilities among glaucoma patients. A combination of visual rehabilitation of low vision therapy and occupational therapy is ideal. Although, there is improvement in reading ability and mobility post low visual aid rehabilitation but there is no evidence on glaucoma patients specifically12. Improvement in daily living and dependency may improve their QoL. Happiness perhaps may improve the balance between oxidative stress damage and antioxidant level. Many previous studies discovered that various biomarkers of oxidative stress are elevated in people with depression, and anxiety disorders13. Similarly, oxidative stress has been implicated in pathogenesis of glaucoma and accelerates retinal ganglion cell damage in glaucoma14. Indirectly, improvement of QoL will help in halting the progression of visual field defect. Based on the previous research project on Malays in Malaysia, navigation and mobility has been identified to be mostly affect in primary glaucoma patients based on QoL questionnaires. Physical activities have potential protective effect against progression and severity of glaucoma9. Improvement in navigation, physical activities and reading ability, perhaps may improve their QoL. The main problem is how do we improve their navigation, physical activities and reading ability despite their constricted visual field. The most important step is to understand the problem and issues pertaining to the navigation, physical activities and reading faced by patients with glaucoma.

DETAILED DESCRIPTION:
Objectives General objective: to develop, validate and evaluate the effectiveness of navigation, physical activities and reading abilities (the new rehabilitation protocols) in Malay adults with primary glaucoma.

Specific objectives:

1. To identify problems with navigation, physical activities and reading in Malay adults with primary glaucoma
2. To develop and validate the new rehabilitation protocols for patients with primary glaucoma
3. To evaluate the effectiveness of the new rehabilitation protocols in improving the quality of life of primary glaucoma patients
4. To evaluate the mean changes of total antioxidant level pre- and post-intervention with the new rehabilitation protocols in primary glaucoma patients
5. To evaluate the changes of ocular parameters pre- and post-intervention with the new rehabilitation protocols in primary glaucoma patients Research design

This research project will be divided into 3 phases with different research designs:

Phase 1: case control study on factors affecting navigation, physical activities and reading between primary glaucoma patients and age matched controls.

Phase 2: development and validation study on new rehabilitation program for navigation, physical activities and reading.

Phase 3: randomized control trial study to evaluate the effectiveness of rehabilitation program and exercise on clinical parameters, quality of life and oxidative stress of primary glaucoma patients.

Study area

A. Glaucoma clinic for patient recruitment, assessment and follow up in:

Hospital Universiti Sains Malaysia (HUSM), Kota Bharu, Kelantan, Malaysia Hospital Raja Perempuan Zainab II (HRPZII), Kota Bharu, Kelantan, Malaysia Hospital Sultanah Bahiyah (HSB), Alor Setar, Kedah, Malaysia Hospital Melaka, Melaka, Malaysia

B. Occupational rehabilitation, Rehabilitation Unit for visual rehabilitation program in:

Hospital Universiti Sains Malaysia (HUSM) Kota Bharu, Kelantan, Malaysia Hospital Raja Perempuan Zainab II, Kota Bharu, Kelantan, Malaysia Hospital Sultanah Bahiyah, Alor Setar, Kedah, Malaysia Hospital Melaka, Melaka, Malaysia Study population Reference population: Primary glaucoma patients-primary open angle glaucoma (POAG) and primary angle closure glaucoma (PACG) Target population: Primary glaucoma patients (POAG and PACG) who attended glaucoma clinic in HUSM, HRPZII, HSB and Hospital Melaka Source population: Patients aged 40 to 70 years old diagnosed with POAG or PACG who are attending the glaucoma clinic, HUSM, HRPZII, HSB and Hospital Melaka from June 2020 until February 2020.

Sampling frame: Glaucoma database in eye clinic of HUSM, HRPZII, HSB and Hospital Melaka Sampling method and subject recruitment The sampling method is based on the specific objective and phases of the study For objective 1: a simple random sampling will be used. For objective 2: convenience sampling.

For objective 3, 4 and 5: randomized Controlled Trial will be conducted. Using block randomization method with sequentially numbered in opaque sealed envelopes (SNOSE), the eligible patients will be randomized into:

Group A: Intervention group Group B: Non-intervention group Primary investigators (Postgraduate students) will be blinded.

Operational definition Primary Open Angle Glaucoma (POAG): A chronic, progressive optic neuropathies that characterised by structural changes in the optic nerve head and/ or with visual field defect without identifiable causes (Asia Pacific Glaucoma guidelines, 2008).

Primary Angle Closure Glaucoma (PACG): An eye with an occludable drainage angle and features indicating that trabecular obstruction by the peripheral iris has occurred, such as peripheral anterior synechiae, elevated intraocular pressure and optic neuropathy (Foster et al., 2002).

Target Intraocular pressure: Target intraocular pressure throughout this study is dependent on severity of the disease based on threshold IOP (Sihota et al., 2018). In this study, target intraocular pressure will be personalized accordingly.

Lens status: Phakic is defined as patients with an intact natural lens without visually significant cataract. A person with visually significant cataract was defined by having, in either eye: any LOCS II grading of ≥2, best-corrected visual acuity of <6/12 in the cataractous eye, cataract as primary cause of vision impairment in that eye, and patient report that general vision was fair, poor, very poor, or blind (Ritcher et al, 2009). Pseudophakic refers to patients who have underwent lens extraction procedure with implantation of artificial intraocular lens for more than 3 months prior to recruitment.

Compliance to treatment: Patients who adhere and persistent to instillation of topical intraocular pressure lowering medications as recommended by their physician throughout follow up (Robin et al, 2011). Adherence is defined as less than 3 times missed their medication in a week. Persistence is defined as continuously on prescribed medication for more than 3 months.

Visual rehabilitation: The process of treatment and education that helps individuals who are visually disabled to attain maximum function, a sense of wellbeing, a personally satisfying level of independence, and optimum quality of life (American Optometric Association, 2004).

Reading speed: rate at which a person reads written text (printed or electronic) in a specific unit of time (Muñoz B et al, 2000).

In this study, the definition of reading speed will differ according to the task of reading and the reading material.

1. Reading speed in reading the Bahasa Malaysia reading chart: number of words read per minute
2. Reading the newspaper print and pharmacy label print: time taken to finish a reading task in minute
3. Reading book: number of pages read per hour/day Eye movement during reading: movement of the eye between the start of first saccade and the end of final saccade during the reading (Muñoz B et al, 2000).

Head movement during reading: all head movement during reading including of modulatory-velocity component with eye saccades and constant-velocity component independent of eye saccades (Muñoz B et al, 2000).

Quality of life: The term "quality of life (QoL)" is defined by the World Health Organization as individuals' perception of their position in life in the context of culture and value systems in which they live in relation to their goals, expectations, standards and concerns (World Health Group, 1995). Total scoring and each domain score of Bahasa Malaysia version GlauQoL -36 questionnaires will be used to determine the QoL. It has been translated and validated and piloted in 96 samples. All 36 translated questions were retained as the Cronbach alpha was found to be 0.85 (Chandramohan et al, 2015).

Depression: a feeling of depressed mood or loss of interest with at least five out of nine symptoms present for a diagnosis of major depression. The mGDS 14 questionnaire was used in this study to assess depression among primary glaucoma patients.

Bump: body contact above the knee, excluding the hands-on adjacent objects. Stumble: a change in posture or gait due to contact with an object below the knee.

Data collection method

This study will be divided into three phases:

1. Phase 1: identification factor affecting navigation, physical activities & reading
2. Phase 2: development and validation of rehabilitation for navigation, physical activities & reading
3. Phase 3: evaluation of the effectiveness of rehabilitation on clinical parameters, quality of life and oxidative stress Phase 1 A case control study will be conducted involving POAG and PACG patients with different severity according to Esterman binocular visual field. An age-matched control subjects will also be recruited. We estimated a sample size of 40 glaucoma subjects and 40 age-matched controls. Selected patients must be physical and mentally fit. Simple random sampling will be applied to patients who attend ophthalmology clinic for other ophthalmological conditions except for glaucoma especially those who were on follow-up for dry eye, non-visually significant cataract, pseudophakic patients. Patients that fulfil the inclusion and exclusion criteria will be selected during their follow up. These patients will be grouped as controls.

Ocular examination: Baseline examination will be conducted in all subjects including visual acuity assessment, contrast sensitivity, stereoacuity and Esterman binocular visual field.

Navigation & physical activities: A stimulated area will be created using the existing facility in occupation rehabilitation unit, HUSM. Similar set up will be conducted in HRPZII, Hospital Sultanah Bahiyah and Hospital Melaka. Glaucoma patients and age-matched control subjects will be asked to navigate in the stimulated area and several areas will be equipped with closed circuit television (CCTV).

A predefined obstacle course navigation will be used to measure mobility performance among glaucoma and control groups. Subjects will be instructed to walk through the course as quickly and safely as possible while avoiding all obstacles in their path. The course will be constructed in a maze form, 30m length in total and seeded with obstacles made with styrofoam that represent objects in a patient's home environment. The illumination along the path range from 100 to 300 lux. Before walking through the course, participants will be given instructions and directions to ensure that they understood the path.

Mobility performance will be assessed by the time required to complete the obstacle course and the number of mobility incidents, which included bumps, stumbles, and orientation problems. A bump will be defined as a body contact above the knee, excluding the hands. A stumble will be defined as a change in posture or gait due to contact with an object below the knee. An orientation problem will be defined as a change in direction that was not consistent with the instructions. A trained observer will be following the participants closely behind to record time and bumps. Surveillance system comprising video camera to record the activities will be implemented as well. Errors are quantified on a 3 point scale, where errors were scored as 1 point if the subject made contact with an obstacle but was able to correct in ≤ 5 sec, 2 points if the subject took 5-15 sec to correct errors, and 3 points if the subject took > 15 sec to self-correct or required the assistance of one of the research assistants to correct the error. Travel time will be converted into walking speed (meters per second) by dividing the distance of established travel path by the time to complete the course. The converted measure permits a direct comparison of mobility performance across other routes and studies.

Special exercise: A special exercise will be designed that is safe for person with constricted visual field; combination of isometric and aerobic exercise. IOP will be taken at baseline and at certain phases of the exercise. If there is an increase of more than 20% from baseline IOP at certain phase of the exercise, that phase will be excluded or replaced accordingly.

Reading: Subject will be asked to read at 40cm (reading distance) with the reading material on a special pedestal. Reading materials include:

1. Universiti Teknologi Mara -Malay related words (UiTM-MrW)
2. Universiti Teknologi Mara- Malay unrelated words (UiTM-MuW)
3. Different sizes of text of common reading materials (Bahasa Malaysia):

   * Pharmacy label print (0.131° print)
   * Newspaper print size (0.26° print)
   * Small newspaper headline/heading size (0.525° print)
   * Large newspaper headline size (1.71° print)
4. A book in Bahasa Malaysia will be selected Reading speed will be assessed using Matlab version 8.3 programme. Eye and head trackers will be used (Polhemus Visiontrak Desktop 300) to document the head and eye movement. Reading will be done in a fix light intensity (500-600lux). A rehabilitation reading regime with or without low vision aid will be designed.

Phase 2

From phase 1 findings, a special rehabilitation device and programme will be designed for:

1. Navigation and mobility
2. Exercise
3. Reading A user friendly and inexpensive device and program with minimal usage of low vision aid will be designed and piloted for 30 glaucoma patients and 30 controls. Simple random sampling will be applied on the patients and control subjects recruited for phase 1 study. An advertisement is also attached here(phase 2).

Devices will include wearable body sensor vibrator and special smartphone apps for recognition of objects. The control subject will be using the special glasses (available in the department) that simulated constricted visual field. For the pilot study, the effectiveness will be considered based on the evaluation conducted for phase 1. The recruited subjects will be asked to practice according to the rehabilitation protocol for 2 weeks. Improvement will be made based on the outcome of the pilot study.

Validation process:

After development or modification of the program, the recruited subjects will be trained and asked to perform it at home for two weeks. They will be provided with a dairy (to ensure that they have conducted it daily). They will be seen after two weeks and the rehabilitation method will be assessed using specific questionnaire. Tentative questionnaire is attached here.

Navigation and physical activities- Any step of the program will be eliminated from the program if it is deemed dangerous (20% of the subjects reported bumping, stumbling, fall or near fall), difficult to manoeuvre (20% of the subjects have difficulty or expressed difficulty in performing the step) and impractical (20% of the subjects expressed infrequent of performing the step at home). Assessment will be made based on simple questionnaire, which will be made once the rehabilitation program has been developed.

Exercise - IOP will be obtained from the patients before and 10min after performing each important step of the exercise using tonometer. If any step of the exercise cause elevation of IOP of more than 2mmHg from the baseline IOP will be eliminated and replaced (if deem necessary). Patients will also be asked on the feasibility and practicality using the questionnaire.

Reading- if the reading material (book) is found to difficult, the material will be replaced. Any new movement of the eye or head that is scored difficult to manoeuvre or impractical will be removed. A questionnaire with Likert score scoring will be developed after completion of phase 1.

Definition of acceptable rehabilitation regime are as below:

Navigation and physical activities- reduction of at least 40% of bumping or stumbling to objects or fall in simulated area. An increase of 40% of total step per day based on accelerometer.

Exercise - An increase of 30% of based on accelerometer. Reading -An increase of 20% of reading task and reading speed.

Phase 3

A randomized single blinded control trial study will be conducted using the newly developed rehabilitation programme from phase 2. A known case of POAG and PACG patients who are compliance to treatment and follow up will be selected. Patients involved in phase 1 will not be recruited into this study. A total of 300 patients will be involved (100-navigation and mobility, 100- exercise and 100-reading). Based on the most recent reliable Humphrey visual field, only those who has more than 10 degree from fixation using Estermann binocular analysis will be selected. Other selection includes best corrected visual acuity of 6/60 on the better seeing eye, pseudophakic or phakic (without visually significant cataract) and without history of surgical intervention 3 months prior to recruitment. Those with severe hearing impairment, physical disabilities such as stroke, limbs amputation, macular and retinal pathology, and on low vision aids will be excluded. Using block randomization method with sequentially numbered in opaque sealed envelopes (SNOSE), the eligible patients will be randomized into:

Group A: Intervention group Group B: Non-intervention group In both groups, their usual topical treatment will be continued. They will be advised to be compliance to the existing treatment. This study will take 6 months to complete.

Baseline assessment An introductory session will be conducted to all selected subjects. The purpose of the study will be explained, and compliance will be emphasized. Venesection will be conducted and 3cc of blood will be obtained. The blood will be kept in the plain bottles and analysed for the level of total anti-oxidant capacity (TAC).

Patients (in group A & B) will be given the GlauQol-36 and mGDS-14 questionnaire in Bahasa Malaysia (Appendix A & B) and be given adequate time to read and answer the questionnaire. If the patient does not understand the questionnaire, they can obtain clarification from the primary investigators (SMCM & NS). The GlauQoL-36 questionnaire consists of 36 questions grouped into 7 domains (daily life, driving, psychological well-being, self-image, anxiety, burden of treatment and confidence in healthcare). Each question was given 4- and 5- point on the Likert scale. The total score from each domain was summed and the score calculated. The mGDS-14 questionnaire consists of 14 questions. It has a yes/no answer and is scored 1 or 0 for each question. Patients with the score of 8 and above are considered depressed.

Accelerometer will be given to the patients with the instruction to wear it all day long except for sleeping and bathing. A baseline reading speed, visual span, eye and head movement will be obtained in those involved in reading rehabilitation program using the reading charts, newspaper and pharmacy label print. These assessments will be conducted twice; before the rehabilitation program and after 6 months of the program. Reading materials in Bahasa Malaysia (a book to read) will also be given. Clinical parameters including IOP and ONH imaging to assess the RNFL thickness and ONH parameters will also be conducted.

Rehabilitation regime

A.Navigation & mobility:

The rehabilitation sessions will be conducted in the Rehabilitation Medicine Unit of HUSM, HRPZII and Hospital Melaka provided by the Occupational Therapy division. The patient is expected and encouraged to come with a carer (who live together with the patient) during the early part of the sessions. After randomization, patients in the group A will be assessed using modified Barthell index, the patient's limitations in daily activities with special attention to the components related to restricted visual field. An introductory session will be conducted by the occupational rehabilitation therapist (baseline), patients will be asked to practice it at home.

Depending on the respective limitations the patient will be taught of ways to get around the problems, emphasizing on the Visual Perception and Sensory Motor Ability as outlined by the Chessington Occupational Therapy Neurological Assessment Battery to maximize function, health and wellbeing. A set of realistic goals will be established together with the patient whether using the restorative or compensatory methods to promote motivation and enhance confidence. Restorative method includes restorative visual field training, optokinetic training and and search task training focussed at improving the loss in visual field or disability arises from the loss of patient's eye field. Interventions involve compensation which are strategies to minimize mismatch in the patient's ability with task difficulty; and substitution which can include environmental modifications to enhance vision such as adjustment of lighting. Subsequent sessions will involve consolidation of the concepts with supervised practices comprising indoor and outdoor activities to enhance patients' understanding and confidence and encourage participation.

Rehabilitation education and activities include:

1. Dressing Light closet to improve acuity. Hang matching clothes together. Pin socks together when placing them in the washer so they will stay matched.
2. Feeding Provide high contrast. Ensure that plates contrast with table surface. Avoid patterned table clothes. Arrange food on the plate in a clockwise fashion and orient the person to the arrangement.
3. Personal hygiene and grooming activities Reduce clutter in bathroom and kitchen cabinets. Use high contrast bathmat and minified mirrors
4. Communication and environmental hardware adaptations Use talking watches or clocks to tell time and high contrast doorknobs.
5. Functional mobility Mobility is eased with the clearing of pathways and the minimizing of clutter and furniture. Lighting in hallways and entryways is also needed. The person with constricted visual field needs to optimize visual scanning abilities by learning to turn and position the head frequently when mobile or participating in an activity.
6. Scanning activity or search task While focusing on a point central to the visual axis, the patient is asked to arrange wooden cubes forming vertical and horizontal lines one at a time. The instruction will be given to arrange from left to right, then right to left, top to bottom and lastly bottom to the top. Patient's visual field is estimated and described to the patient. Patient is advised on the 'danger area' outside the visual field that can pose various risks to the patient.
7. Room orientation and memory This is applied to a small area such as a bedroom or a toilet. The patient is asked to stand inside a simulated room in the Rehabilitation Unit and describe the names of the objects that he/she can see. Emphasizing on the location of the objects and their directions from the patient (right, left, in front, behind), patient is trained to systematically orientate himself in the room relative to those objects. Certain objects are highlighted to the patient as a precaution to avoid stumbles and falls. For safety, cleaning supplies should be placed separately from food supplies.
8. Orientation and mobility This activity covers a larger area that the patient will be in which is the patient's home. Patient will be instructed regarding room familiarisation according to the house's structure as described by patient's carer with the help of a drawing. For example, the patient is taught to memorize the number of steps needed to be made to get to the toilet from his room, and in what direction.
9. Reading (this is not part of the reading rehabilitation) Patient will be taught to label the things that are of importance to them at home to aid recognition, for example bottles of spice. The letters should be of appropriate size deemed legible by the patient according to the patient's field of view, and of high contrast. For patients on medications, they are advised to use medication organizer to get them organized.
10. Eye-hand coordination To enhance hand-eye coordination, a pegboard is used as a form of exercise for the patient. Patient is asked to match coloured pegs into its corresponding holes according to a reference template. This training also allows the patient to get used to the extent of field of view that he possesses.
11. Optokinetic training programme This programme is built based on the knowledge that eye and body movements are coordinated by the same parts of the brain, which is important in maintaining stability and balance. Repeated training helps to re-teach the body of its responsible actions, by the means of precise eye movements. This is done via optokinetic eye programme to accelerate physical and mental fitness. Fortunately, the high functional adaptability of the brain permits positive training and learning as the person ages.

Occupational therapist will conduct a home visit if necessary. A diary will be given to assess their compliance. Reassessment will be done for every 2 weeks for 2 months and every month for the next 2 months. Another home visit will be conducted if the patients show poor understanding or compliance during the re-assessment evaluation.

Patients in group B will also be given a diary to record their activities. In both groups, their usual topical treatment will be continued. They will be advised to be compliance to the existing treatment.

B. Special exercise:

An instruction course will be conducted and a CD (with step by step exercise demonstration) will be given to the patients in group A. They will be asked to come for another session in 2 weeks. Then they will be asked to conduct the exercise for at least three times a week. Exercise diary and accelerometer will also be given to patients of both groups.

C. Reading regime:

A briefing will be given to all the patients involved in this regime. Patients in both groups will be asked to complete a reading task (reading the given book) a day; number of pages completed in an hour per day, and time taken to complete a page in the given book. They will be asked to record the time they have completed the task in their reading diary. Any extra reading task will also be recorded this include reading Quran and newspaper.

Final assessment At 6 months post recruitment, patients in group A and B will be asked to complete the Malay version of Glau-QOL 36 and MGD14. Accelerometer reading will also be documented. The number of pages read for the given task will be compiled. The reading diary will be evaluated. Reading speed will be calculated daily and the mean reading speed will be used for analysis. Another venesection will be conducted to examine the level of TAC. Clinical assessment including IOP, RNFL thickness and ONH parameters will be conducted.

Serum TAC analysis Level of TAC analysis will be conducted using using QuantiChromTM Antioxidant Assay Kit (DTAC-100). It will be centrifuged 10 min at 14000 rpm, the plasma will be used as sample for calculation of total antioxidant capacity (TAC). Plasma can be stored in a freeze at -80°C in the laboratory (stable for 1 month) for future analysis if required. After preparing the reagent provided from the test kit (DTAC-100), patient plasma will be mixed with the diluted reagent in a plate which will be read at optical density of 570nm. The result obtained will be plotted against the standard concentration and a standard curve is obtained. By using the graph plotted and a formula provided in the test kit, the serum TAC will be calculated. Serum total antioxidant capacity will be calculated at baseline and at six months post recruitment.

Data Entry and Statistical Analysis The data entry and analysis will be performed by using Statistical Package for the Social Sciences (SPSS) version 22 licensed to USM. For numerical data, paired t-test will be used to compare the changes at baseline and 6 months post intervention. Multivariate analysis will also be conducted

ELIGIBILITY:
Inclusion Criteria:

1. Known cases of POAG and PACG who are compliance to treatment and follow up
2. Those who have more than 10 degree from fixation (based on Humphrey visual field)
3. Best corrected visual acuity of 6/60 on the better seeing eye
4. Pseudophakic or phakic (without visually significant cataract)

Exclusion Criteria:

1. History of surgical intervention 3 months prior to recruitment
2. Physical disabilities such as stroke, limbs amputation
3. Severe hearing impairment
4. Those with macular and retinal pathology
5. Those already on low vision aids

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Navigation: completion of maze | Baseline (before randomization)
  Time to complete the maze (minutes)
Navigation: completion of maze | 24 weeks after randomization
  Time to complete the maze (minutes)
Navigation: number of obstacles | Baseline (before randomization)
  Number of stumbles and bumps while walking through the maze (number)
Navigation: number of obstacles | 24 weeks after randomization
  Number of stumbles and bumps while walking through the maze (number)
Mobility at home | Baseline (before randomization)
  Accelerometer reading (steps/day)
Mobility at home | 2 weeks after randomization
  Accelerometer reading (steps/day)
Mobility at home | 4 weeks after randomization
  Accelerometer reading (steps/day)
Mobility at home | 8 weeks after randomization
  Accelerometer reading (steps/day)
Mobility at home | 16 weeks after randomization
  Accelerometer reading (steps/day)
Mobility at home | 24 weeks after randomization
  Accelerometer reading (steps/day)
Physical activity and exercise | Baseline (before randomization)
  Accelerometer reading of moderate-vigorous physical activity (MVPA) (number)
Physical activity and exercise | 2 weeks after randomization
  Accelerometer reading of moderate-vigorous physical activity (MVPA) (number)
Physical activity and exercise | 4 weeks after randomization
  Accelerometer reading of moderate-vigorous physical activity (MVPA) (number)
Physical activity and exercise | 8 weeks after randomization
  Accelerometer reading of moderate-vigorous physical activity (MVPA) (number)
Physical activity and exercise | 16 weeks after randomization
  Accelerometer reading of moderate-vigorous physical activity (MVPA) (number)
Physical activity and exercise | 24 weeks after randomization
  Accelerometer reading of moderate-vigorous physical activity (MVPA) (number)
Reading speed of near vision chart | Baseline (before randomization
  Number of words per minute
Reading speed of near vision chart | 24 weeks after randomization
  Number of words per minute
Reading speed of the provided materials (prescription label and newspaper) | Baseline (before randomization)
  Number of words per minute
Reading speed of the provided materials (prescription label and newspaper) | 24 weeks after randomization
  Number of words per minute
Reading speed of the given book | Baseline (before randomization)
  Number of pages per hour
Reading speed of the given book | 8 weeks after randomization
  Number of pages per hour
Reading speed of the given book | 16 weeks after randomization
  Number of pages per hour
Reading speed of the given book | 24 weeks after randomization
  Number of pages per hour
Quality of life score | Baseline (before randomization)
  Total score from each domains of Bahasa Malaysia version of Glaucoma Quality of life 36 questionnaire (GlauQoL 36) using likert scoring 1-5
Quality of life score | 24 weeks after randomization
  Total score from each domains of Bahasa Malaysia version of Glaucoma Quality of life 36 questionnaire (GlauQoL 36) using likert scoring 1-5
Depression score | Baseline (before randomization)
  Using Bahasa Malaysia version of geriatric depression scale 14 (MGDS 14) questionnaire.
  The score of 8 and above is considered as depressed.
Depression score | 24 weeks after randomization
  Using Bahasa Malaysia version of geriatric depression scale 14 (MGDS 14) questionnaire.
  The score of 8 and above is considered as depressed.
Serum total anti-oxidant capacity (TAC) | Baseline (before randomization)
  The concentration of the TAC level (Ta) using a commercialized kit (QuantiChromTM Antioxidant Assay Kit (DTAC-100, BioAssay System, USA)
Serum total anti-oxidant capacity (TAC) | 24 weeks after randomization
  The concentration of the TAC level (Ta) using a commercialized kit (QuantiChromTM Antioxidant Assay Kit (DTAC-100, BioAssay System, USA)

SECONDARY OUTCOMES:
Intraocular pressure (IOP) | Baseline (before randomization)
  Measurement of intraocular pressure (mmHg) using Goldman Applanation Tonometry(Haag-Street International, UK)
Intraocular pressure (IOP) | 8 weeks after randomization
  Measurement of intraocular pressure (mmHg) using Goldman Applanation Tonometry(Haag-Street International, UK)
Intraocular pressure (IOP) | 16 weeks after randomization
  Measurement of intraocular pressure (mmHg) using Goldman Applanation Tonometry(Haag-Street International, UK)
Intraocular pressure (IOP) | 24 weeks after randomization
  Measurement of intraocular pressure (mmHg) using Goldman Applanation Tonometry(Haag-Street International, UK)
Retinal nerve fiber layer thickness (RNFL) | Baseline (before randomization)
  Measurement of RNFL thickness (mm) using HD Cirrus Optical Coherent Tomography (Carl Zeiss) Mesurement of RNFL thickness using HD Cirrus Optical Coherent Tomography (Carl Zeiss, US)
Retinal nerve fiber layer thickness (RNFL) | 8 weeks after randomization
  Measurement of RNFL thickness (mm) using HD Cirrus Optical Coherent Tomography (Carl Zeiss) Mesurement of RNFL thickness using HD Cirrus Optical Coherent Tomography (Carl Zeiss, US)
Retinal nerve fiber layer thickness (RNFL) | 24 weeks after randomization
  Measurement of RNFL thickness (mm) using HD Cirrus Optical Coherent Tomography (Carl Zeiss) Mesurement of RNFL thickness using HD Cirrus Optical Coherent Tomography (Carl Zeiss, US)

CONTACTS AND LOCATIONS:
Overall Officials: Liza Sharmini Ahmad Tajudin, Prof. Dr., Principal Investigator — Department of Ophthalmology, School of Medical Sciences, Universiti Sains Malaysia
Locations (1):
- Universiti Sains Malaysia, Kota Bharu, Kelantan, Malaysia

REFERENCES:
- [Result] Tham YC, Li X, Wong TY, Quigley HA, Aung T, Cheng CY. Global prevalence of glaucoma and projections of glaucoma burden through 2040: a systematic review and meta-analysis. Ophthalmology. 2014 Nov;121(11):2081-90. doi: 10.1016/j.ophtha.2014.05.013. Epub 2014 Jun 26. PMID 24974815
- [Result] Weinreb RN, Aung T, Medeiros FA. The pathophysiology and treatment of glaucoma: a review. JAMA. 2014 May 14;311(18):1901-11. doi: 10.1001/jama.2014.3192. PMID 24825645
- [Result] Friedman DS, Freeman E, Munoz B, Jampel HD, West SK. Glaucoma and mobility performance: the Salisbury Eye Evaluation Project. Ophthalmology. 2007 Dec;114(12):2232-7. doi: 10.1016/j.ophtha.2007.02.001. Epub 2007 Nov 5. PMID 17980433
- [Result] Turano KA, Rubin GS, Quigley HA. Mobility performance in glaucoma. Invest Ophthalmol Vis Sci. 1999 Nov;40(12):2803-9. PMID 10549639
- [Result] Viswanathan AC, McNaught AI, Poinoosawmy D, Fontana L, Crabb DP, Fitzke FW, Hitchings RA. Severity and stability of glaucoma: patient perception compared with objective measurement. Arch Ophthalmol. 1999 Apr;117(4):450-4. doi: 10.1001/archopht.117.4.450. PMID 10206571
- [Result] Izzotti A, Bagnis A, Sacca SC. The role of oxidative stress in glaucoma. Mutat Res. 2006 Mar;612(2):105-14. doi: 10.1016/j.mrrev.2005.11.001. Epub 2006 Jan 18. PMID 16413223
- [Result] Majsterek I, Malinowska K, Stanczyk M, Kowalski M, Blaszczyk J, Kurowska AK, Kaminska A, Szaflik J, Szaflik JP. Evaluation of oxidative stress markers in pathogenesis of primary open-angle glaucoma. Exp Mol Pathol. 2011 Apr;90(2):231-7. doi: 10.1016/j.yexmp.2011.01.001. Epub 2011 Jan 15. PMID 21241689
- [Result] Markowitz M. Occupational therapy interventions in low vision rehabilitation. Can J Ophthalmol. 2006 Jun;41(3):340-7. doi: 10.1139/I06-020. PMID 16767190
- [Result] McKean-Cowdin R, Wang Y, Wu J, Azen SP, Varma R; Los Angeles Latino Eye Study Group. Impact of visual field loss on health-related quality of life in glaucoma: the Los Angeles Latino Eye Study. Ophthalmology. 2008 Jun;115(6):941-948.e1. doi: 10.1016/j.ophtha.2007.08.037. Epub 2007 Nov 12. PMID 17997485
- [Result] Nilsson UL. Visual rehabilitation of patients with advanced stages of glaucoma, optic atrophy, myopia or retinitis pigmentosa. Doc Ophthalmol. 1988 Dec;70(4):363-83. doi: 10.1007/BF00157066. PMID 3266961
- [Result] Chong Seong NT, Yaakub A, Jalil RA, Tirmandas Vn K, A/P Sandragasu T, Noor JBM, Husain NB, Mustari ZB, Hamid SAA, Mt Saad AB, At LS. Effect of physical activity on severity of primary angle closure glaucoma. Ther Adv Ophthalmol. 2019 Jul 29;11:2515841419864855. doi: 10.1177/2515841419864855. eCollection 2019 Jan-Dec. PMID 31384724
- [Result] Ramulu PY, Maul E, Hochberg C, Chan ES, Ferrucci L, Friedman DS. Real-world assessment of physical activity in glaucoma using an accelerometer. Ophthalmology. 2012 Jun;119(6):1159-66. doi: 10.1016/j.ophtha.2012.01.013. Epub 2012 Mar 2. PMID 22386950
- [Result] Ramulu P. Glaucoma and disability: which tasks are affected, and at what stage of disease? Curr Opin Ophthalmol. 2009 Mar;20(2):92-8. doi: 10.1097/ICU.0b013e32832401a9. PMID 19240541
- [Result] Ramulu PY, West SK, Munoz B, Jampel HD, Friedman DS. Glaucoma and reading speed: the Salisbury Eye Evaluation project. Arch Ophthalmol. 2009 Jan;127(1):82-7. doi: 10.1001/archophthalmol.2008.523. PMID 19139345
- [Result] Sacca SC, Izzotti A, Rossi P, Traverso C. Glaucomatous outflow pathway and oxidative stress. Exp Eye Res. 2007 Mar;84(3):389-99. doi: 10.1016/j.exer.2006.10.008. Epub 2006 Dec 29. PMID 17196589
- [Result] Salim S. Oxidative stress and psychological disorders. Curr Neuropharmacol. 2014 Mar;12(2):140-7. doi: 10.2174/1570159X11666131120230309. PMID 24669208
- [Result] Stelmack JA, Tang XC, Wei Y, Wilcox DT, Morand T, Brahm K, Sayers S, Massof RW; LOVIT II Study Group. Outcomes of the Veterans Affairs Low Vision Intervention Trial II (LOVIT II): A Randomized Clinical Trial. JAMA Ophthalmol. 2017 Feb 1;135(2):96-104. doi: 10.1001/jamaophthalmol.2016.4742. PMID 27978569
- [Result] van Landingham SW, Willis JR, Vitale S, Ramulu PY. Visual field loss and accelerometer-measured physical activity in the United States. Ophthalmology. 2012 Dec;119(12):2486-92. doi: 10.1016/j.ophtha.2012.06.034. Epub 2012 Aug 11. PMID 22892152
- [Result] Wilkinson ME, Shahid KS. Low vision rehabilitation: An update. Saudi J Ophthalmol. 2018 Apr-Jun;32(2):134-138. doi: 10.1016/j.sjopt.2017.10.005. Epub 2017 Oct 27. PMID 29942183